CLINICAL TRIAL: NCT01638962
Title: The Effect on Knee Joint Loads of Instruction in Analgesic Use Compared With NEUROMUSCULAR Exercise in Patients With Knee Osteoarthritis - A Single Blind RCT
Brief Title: The Effect on Knee Joint Loads of Analgesic Use Compared With Exercise in Patients With Knee Osteoarthritis - An RCT
Acronym: EXERPHARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Region Syddanmark (Other); The Danish Rheumatism Association (Other); Association of Danish Physiotherapists (Other)
Responsible Party: Principal Investigator, Brian Clausen, PT, PhD-student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20110153
Record Dates: First submitted 2012-07-03; First posted 2012-07-12 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Exercise Therapy; Gait; Joint load; Knee Joint; Middle Aged; Osteoarthritis, Knee/therapy; Pain Management
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Agnosia | interventions — Analgesia; Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen; Aspirin; Celecoxib; dexibuprofen; Etoricoxib; lornoxicam; Meloxicam; Diclofenac; Etodolac; Indomethacin; Nabumetone; Naproxen; tenoxicam; tiaprofenic acid; dexketoprofen trometamol; Muscle Stretching Exercises; Exercise; Functional Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEMEX (Experimental): NEuroMuscular EXercise
  Interventions: Other: Neuromuscular exercise
- PHARMA (Active Comparator): PHARMAcological pain relief
  Interventions: Drug: Instruction on analgesic use for pain relief (acetaminophen and NSAIDs)

INTERVENTIONS:
Drug: Instruction on analgesic use for pain relief (acetaminophen and NSAIDs) — The PHARMA group receives instruction, by video and pamphlet, on how to best use acetaminophen and NSAID as pain management for knee OA.
  Other Names: Acetaminophen; Non-Steroid Anti-Inflamatoric Drug:; Ibuprofen; Acetylsalicylic acid; Celecoxib; Dexibuprofen; Etoricoxib; Lornoxicam; Meloxicam; Diclofenac; Etodolac; Indomethacin; Nabumetone; Naproxen; Tenoxicam; Tiaprofenic acid; Dexketoprofen
  Arms: PHARMA
Other: Neuromuscular exercise — The exercise group receives 1 hour of supervised neuromuscular exercise two times a week for 8 weeks. Supervision is conducted by physiotherapists specially trained in using neuromuscular exercise and its principles.
  Other Names: Exercise; Stability; Alignment; Functional
  Arms: NEMEX

SUMMARY:
The purpose of this study is to compare the effects of neuromuscular exercise and analgesic use on knee joint load, in patients with mild to moderate knee osteoarthritis (OA).

It is expected that the two groups will receive equipotent pain relieving effect, despite this, the investigators expect a between group difference in knee joint load, and the exercise group will have a reduction in knee joint load.

ELIGIBILITY:
Inclusion Criteria:

* Compliance with the ACR criteria
* Medial knee OA defined as "No osteoarthritis", "Doubtful narrowing of joint space and/or possible osteophytes", "Definite osteophytes and possible narrowing of joint space", "Multiple osteophytes, definite narrowing of joint space and some sclerosis and deformity of bone ends". This corresponds to the Kellgren and Lawrence (KL) grades 0, 1, 2 and 3 respectively
* Willingness to participate in exercise and use of analgesics
* A maximum of 75/100 points in the KOOS Pain subscale
* BMI of 32 or less

Exclusion Criteria:

* Medial greater than lateral joint space width
* Medial knee OA of KL grade 4
* Knee surgery or steroid injection within the past 6 months
* Already taking max dose NSAIDs or acetaminophen
* Any physician-determined condition that is a contraindication for use of acetaminophen, NSAIDs or to exercise
* Problems affecting the lower extremity overriding the problems from the knee
* Knee surgery planned in the next 6 months
* Known ACL tear within the past 6 months
* ACL reconstruction
* Diagnosis of systemic arthritis
* Difficulty complying with treatment schedule
* Inability to fill out questionnaires
* Inability to ambulate without an assistive device
* Ankle, knee or hip replacement
* Tibial/femoral osteotomy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 1st peak RMS (root mean square) Knee Index. | Baseline and post intervention (8 weeks)
  1st peak RMS Knee Index, is combined of the moments of the 3 planes working over the the knee; flexion, adduction and internal rotation moments. Measured with the Vicon system.
  1st peak RMS knee moment = √(Kflex. moment2 + Kadd. moment2 + Kint.rot. moment2 )/3

SECONDARY OUTCOMES:
Change from baseline in 1st peak Knee adduction moment | Baseline and post intervention (8 weeks)
Change from baseline in the KOOS (Knee injury and Osteoarthritis Outcome Score) questionnaire | Baseline and post intervention (8 weeks)
Change from baseline in Maximum number of one-leg rises from stool test | Baseline and post intervention (8 weeks)
  This test evaluates maximal performance and muscle strength in the lower extremity
Change from baseline in Maximum number of knee-bendings in 30s test | Baseline and post intervention (8 weeks)
  This test evaluates the ability to perform fast changes between eccentric and concentric muscle force over the knee joint
Change from baseline in One-leg hop for distance test | Baseline and post intervention (8 weeks)
  The test mimics sporting activities and demands muscle explosivety, balance and functional stability of the knee

CONTACTS AND LOCATIONS:
Overall Officials: Brian Clausen, PT, M.Sc., Principal Investigator — Musculoskeletal Function and Physiotherapy, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark; Ewa M. Roos, Professor, Study Chair — Musculoskeletal Function and Physiotherapy, Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Region Syddanmark, Denmark

REFERENCES:
- [Background] Thorstensson CA, Henriksson M, von Porat A, Sjodahl C, Roos EM. The effect of eight weeks of exercise on knee adduction moment in early knee osteoarthritis--a pilot study. Osteoarthritis Cartilage. 2007 Oct;15(10):1163-70. doi: 10.1016/j.joca.2007.03.012. Epub 2007 Apr 26. PMID 17466541
- [Background] Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. BMC Musculoskelet Disord. 2010 Jun 17;11:126. doi: 10.1186/1471-2474-11-126. PMID 20565735
- [Derived] Holsgaard-Larsen A, Christensen R, Clausen B, Sondergaard J, Andriacchi TP, Roos EM. One year effectiveness of neuromuscular exercise compared with instruction in analgesic use on knee function in patients with early knee osteoarthritis: the EXERPHARMA randomized trial. Osteoarthritis Cartilage. 2018 Jan;26(1):28-33. doi: 10.1016/j.joca.2017.10.015. Epub 2017 Oct 26. PMID 29107059
- [Derived] Holsgaard-Larsen A, Clausen B, Sondergaard J, Christensen R, Andriacchi TP, Roos EM. The effect of instruction in analgesic use compared with neuromuscular exercise on knee-joint load in patients with knee osteoarthritis: a randomized, single-blind, controlled trial. Osteoarthritis Cartilage. 2017 Apr;25(4):470-480. doi: 10.1016/j.joca.2016.10.022. Epub 2016 Nov 9. PMID 27836677
- [Derived] Clausen B, Holsgaard-Larsen A, Sondergaard J, Christensen R, Andriacchi TP, Roos EM. The effect on knee-joint load of instruction in analgesic use compared with neuromuscular exercise in patients with knee osteoarthritis: study protocol for a randomized, single-blind, controlled trial (the EXERPHARMA trial). Trials. 2014 Nov 15;15:444. doi: 10.1186/1745-6215-15-444. PMID 25399048